CLINICAL TRIAL: NCT02398825
Title: Optimizing Ponatinib USe (OPUS). A GIMEMA Phase 2 Study of the Activity and Risk Profile of Ponatinib, 30 mg Once Daily, in Chronic Myeloid Leukemia (CML) Chronic Phase (CP) Patients Resistant to Imatinib
Brief Title: Activity and Risk Profile of Ponatinib in Chronic Phase Patients With Chronic Myeloid Leukemia Resistant to Imatinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML1315; 2015-001102-34 (EudraCT Number)
Record Dates: First submitted 2015-03-15; First posted 2015-03-26 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Myeloid Leukemia; Chronic Phase; Adults
Keywords: Chronic myeloid leukemia; Chronic phase; Adults; Ponatinib; Imatinib resistant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ponatinib (Experimental)
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib is given orally 30 mg daily, with dose adjustment to 15 mg daily once a BCR-ABL1 level minor or equal to 0.1% (MMR) has been achieved and confirmed in the next test, 4 weeks apart. A return to prior, 30 mg, dose is due in case of return of BCR-ABL1 transcripts level to > 1%. Dose adjustments for toxicity are detailed in the protocol.

SUMMARY:
This study aims at evaluating the efficacy of treatment with ponatinib in patients with chronic myeloid leukemia who are in a chronic phase and who previously received treatment with imatinib but resulted to be resistant to it.

DETAILED DESCRIPTION:
Phase 2, single-arm, multicentre, open label. No interim analysis is planned, but a monitoring committee will evaluate the data every 6 months. Ponatinib is given orally 30 mg daily, with dose adjustment to 15 mg daily once a BCR-ABL1 level smaller or equal to 0.1% (MMR) has been achieved and confirmed in the next test, 4 weeks apart. A return to prior, 30 mg, dose is due in case of return of BCR-ABL1 transcripts level to > 1%. Dose adjustments for toxicity are detailed in the protocol. Treatment time will be 52 weeks, during which study drug will be provided free-of-charge by ARIAD Pharmaceuticals, upon approval of the protocol. Treatment is discontinued at any time in case of failure or treatment-related SAEs. After one year of treatment, upon request of the local investigator and upon confirmation of the Treatment Advisory Committee (TAC, see section 23), ARIAD Pharmaceutics, Inc. will continue to provide ponatinib for the study patients who will benefit from treatment continuation, for at least 2 years, until the drug will be approved with that indication.

ELIGIBILITY:
Inclusion Criteria:

1. Cytogenetic and/or molecular confirmed diagnosis of Ph+ and/or BCR-ABL1+ CML
2. Age ≥ 18 years
3. Chronic phase CML
4. Prior treatment with imatinib, any dose
5. Resistance to imatinib, as defined by any one of the ELN 2013 failure criteria, as follows:

   * no complete hematologic response (CHR) at 3 months
   * no cytogenetic response (CyR) (Ph+ > 95%) at 3 months
   * Less than partial CyR (PCyR, Ph+ > 35%) at 6 months
   * BCR-ABL1 > 10% at 6 months
   * Non complete CyR (CCyR) (Ph+ > 0%) at 12 months
   * BCR-ABL1 > 1% at 12 months
   * Loss of CHR, at any time
   * Loss of CCyR, at any time
   * Confirmed loss of major molecular response (MMR) (BCR-ABL1 bigger or equal to 0.1% in two consecutive tests, of which one bigger or equal to 1%), at any time
   * Any new BCR-ABL1 mutation, at any time
6. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment
7. An effective form of contraception with their sexual partners from enrolment through 4 months after the end of treatment
8. Signed written informed consent according to ICH/EU/GCP and national local laws prior to any study procedures
9. Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Accelerated or blastic phase CML
2. Patients previously treated with nilotinib or dasatinib
3. Patients with the T315I mutation
4. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis or of alcohol abuse
5. Patients with history of acute myocardial infarction (AMI), unstable angina or coronary heart disease (CHD), congestive heart failure, cerebrovascular events (CVE) (stroke or transitory ischemic attack), or peripheral artery occlusive disease (PAOD)
6. Compelled to take medications that are known to be associated with Torsades de Pointes and/or with significant QTc prolongation
7. Pregnant or breastfeeding
8. Any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the drug
9. Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Number of patients with major cytogenetic response | After 52 weeks of ponatinib treatment start
  Cytogenetic response (CyR) is defined based on the percentage of Ph pos metaphases, as evaluated by chromosome banding analysis (CBA) of at least 20 marrow cell metaphases:
  1. Major Cytogenetic Response if Ph pos metaphases < 35%
  2. Complete (CCyR) if Ph pos metaphases 0 or FISH BCR-ABL1 nuclei minor or equal to 1%
  3. Partial (PCyR) if Ph pos metaphases 1-34%
  4. Minor (mCyR) if Ph pos metaphases 35-65%
  5. Minimal or none (min/none CyR) if Ph pos metaphases > 65% If marrow cell metaphases cannot be obtained or analysed, interphase fluorescence-in-situ-hybridization (FISH) can be used, but only to distinguish a CCyR (minor or equal to 1% positive nuclei out of at least 200 nuclei) from a non CCyR. FISH data cannot be used to classify a response as minimal, minor, or partial.

SECONDARY OUTCOMES:
Number of Cardiovascular Adverse Events (AEs) | After three years from ponatinib treatment start
Number of blood hypertension AEs | After three years from ponatinib treatment start
Number of pancreatitis AEs | After three years from ponatinib treatment start
Number of patients achieving Complete Cytogenetic Response (CCyR) | After 52 weeks of ponatinib treatment start
Number of patients achieving major molecular response | After 52 weeks of ponatinib treatment start
Number of patients with failure-free survival | At 36 months from ponatinib treatment start
Number of patients with progression-free survival | At 36 months from ponatinib treatment start
Number of patients in overal survival | At 36 months from ponatinib treatment start
Number of patients in event-free survival | At 36 months from ponatinib treatment start
Quality of Life patterns over time with the EORTC QLQ-C30 and the EORTC QLQ-CML24 questionnaires | At baseline and at at weeks 4, 12, 24, 36 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Castagnetti, Study Chair — Department of Hematology, S. Orsola-Malpighi University of Bologna
Locations (37):
- Italy (37):
  - Aos Ss. Antonio E Biagio E C. Arrigo - Soc Ematologia, Alessandria
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Sc Ematologia E Ctmo, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo, Catania
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Ao Di Catanzaro "Pugliese-Ciaccio", Presidio Ospedaliero "Ciaccio - de Lellis" - Ematologia, Catanzaro
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Aso S. Croce E Carle - Cuneo - Sc Ematologia, Cuneo
  - Irccs Aou San Martino - Genova - Uo Clinica Ematologica, Genova
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - .R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - Aou Policlinico "G. Martino" - Messina - Uoc Ematologia, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Milano Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Ausl Della Romagna, Ospedale "Santa Maria Delle Croci" - Ravenna - Ematologia, Ravenna
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Ao San Camillo Forlanini - Roma - Uoc Ematologia E Trapianto Cellule Staminali, Roma
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Roma Uoc Pronto Soccorso E Accettazione Ematologica - Dipartimento Biotecnologie Cellulari Ed Ematologia - Università Degli Studi Di Roma "Sapienza", Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Ao S. Maria - Terni - Sc Onco Ematologia, Terni
  - Unità Operativa Di Ematologia - Presidio Ospedaliero Di Treviso - Azienda Ulss N.2 Marca Trevigiana, Treviso
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

REFERENCES:
- See also: GIMEMA Foundation — http://www.gimema.it